CLINICAL TRIAL: NCT00022438
Title: Immunization of HLA-0201 Positive Patients With Metastatic Melanoma Using a Peptide From Tyrosinase-related Protein 2 (TRP-2)
Brief Title: Vaccine Therapy With or Without Interleukin-2 in Treating Patients With Metastatic Melanoma That Has Not Responded to Previous Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068818; NCI-01-C-0193; NCI-5369; NCT00017849 (obsolete NCT alias)
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2004-07

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; incomplete Freund's adjuvant; dopachrome isomerase

INTERVENTIONS:
Biological: aldesleukin
Biological: incomplete Freund's adjuvant
Biological: recombinant tyrosinase-related protein-2

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill tumor cells. Combining vaccine therapy with interleukin-2 may be an effective treatment for metastatic melanoma.

PURPOSE: Randomized phase II trial to compare the effectiveness of vaccine therapy plus interleukin-2 to that of vaccine therapy alone in treating patients who have metastatic melanoma that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical responses in patients with HLA-A0201-positive refractory metastatic melanoma treated with tyrosinase-related protein-2:180-188 peptide vaccine alone.
* Determine the clinical response rate of patients who have an immediate need to receive interleukin-2 (IL-2) in addition to this vaccine.
* Compare the immunologic response, in terms of changes in T-cell precursors before and after treatment, in patients treated with this vaccine with or without IL-2.
* Compare the toxicity profile of these regimens in these patients.

OUTLINE: This is a randomized, open-label study.

Patients who need immediate interleukin-2 (IL-2) receive tyrosinase-related protein-2 (TRP-2):180-188 peptide vaccine emulsified with Montanide ISA-51 on day 1 and high-dose IL-2 IV over 15 minutes once every 8 hours on days 2-5. Treatment repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients who do not need immediate IL-2 are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive TRP-2:180-188 peptide vaccine emulsified with Montanide ISA-51 subcutaneously (SC) on day 1. Treatment repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive TRP-2:180-188 peptide vaccine emulsified with Montanide ISA-51 SC once weekly on weeks 1-4. Treatment repeats every 7 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients who have a complete response (CR) receive 1 additional course after achieving CR. Patients who have progressive disease while receiving vaccine alone may cross over to receive peptide vaccine with IL-2 for at least 2 courses.

Patients are followed at 3 weeks.

PROJECTED ACCRUAL: A maximum of 83 patients (19-33 who need immediate interleukin-2 (IL-2); 15-25 per treatment arm who do not need immediate IL-2) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic melanoma

  * Refractory to standard therapy
  * No resectable locoregional disease
* HLA-A0201 positive
* Measurable disease
* Previously resected brain metastases, brain metastases stable after prior radiosurgery, or brain metastases less than 1 cm and without edema allowed

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 90,000/mm^3
* No coagulation disorders

Hepatic:

* Bilirubin no greater than 2.0 mg/dL (3.0 mg/dL for patients with Gilbert's syndrome)
* AST/ALT less than 3 times normal
* Hepatitis B surface antigen negative

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No major medical illness of the cardiovascular system
* No cardiac ischemia*
* No myocardial infarction*
* No cardiac arrhythmias* NOTE: * For interleukin-2 (IL-2) administration

Pulmonary:

* No major medical illness of the respiratory system
* No obstructive or restrictive pulmonary disease (for IL-2 administration)

Immunologic:

* HIV negative
* No primary or secondary immunodeficiency
* No known immunodeficiency disease
* No autoimmune disease
* No active systemic infections

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic therapy for melanoma
* No prior immunization to tyrosinase-related protein-2 antigen
* No other concurrent biologic therapy for melanoma

Chemotherapy:

* At least 3 weeks since prior chemotherapy for melanoma and recovered
* No concurrent chemotherapy for melanoma

Endocrine therapy:

* At least 3 weeks since prior endocrine therapy for melanoma
* No concurrent systemic steroid therapy
* No concurrent endocrine therapy for melanoma

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy for melanoma and recovered
* No concurrent radiotherapy for melanoma

Surgery:

* See Disease Characteristics

Other:

* No other concurrent therapy for melanoma

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-06; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States